CLINICAL TRIAL: NCT03696966
Title: KU Alternate Meal Energy Level Study
Acronym: KAMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Debra K. Sullivan, PhD, RD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_STUDY00141322
Record Dates: First submitted 2018-09-26; First posted 2018-10-05 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Weight Loss
Keywords: weight management; obesity; very-low calorie diet; intermittent diet
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Calorie Restriction (Active Comparator): Daily calorie restriction: follow low-calorie diet (1,200-1,500 calories) daily using portion-controlled meals
  Interventions: Dietary Supplement: Portion-Controlled Meals; Behavioral: Low-Calorie Diet
- Intermittent Very-Low Calorie Diet (Experimental): Intermittent Restriction: follow very-low calorie diet (500-800) with portion-controlled meals three days per week and structured healthy eating on other days
  Interventions: Dietary Supplement: Portion-Controlled Meals; Behavioral: Intermittent Very-Low Calorie Diet

INTERVENTIONS:
Dietary Supplement: Portion-Controlled Meals — Increase dietary structure using portion-controlled meals (PCM)
Behavioral: Low-Calorie Diet — Restrict calorie intake daily
  Arms: Continuous Calorie Restriction
Behavioral: Intermittent Very-Low Calorie Diet — Severely restrict calorie intake intermittently
  Other Names: Intermittent Fasting
  Arms: Intermittent Very-Low Calorie Diet

SUMMARY:
Compare intermittent versus continuous calorie restriction to learn more about these eating plans and determine whether they are useful and effective to lose weight and keep it off.

DETAILED DESCRIPTION:
The purpose of this study is to provide evidence for the feasibility of an alternative weight control strategy by comparing two diets to see how intermittent calorie restriction compares to continuous or daily calorie restriction for weight loss in 35 adults with overweight or obesity. These diets will be incorporated into a comprehensive and intensive weight management program involving weekly health education meetings, regular diet and physical activity tracking, and feedback from a registered dietitian.

Each intervention includes 3 months of weight loss and 3 months of weight maintenance.

Group 1: Follow a low-calorie diet every day (1,200 - 1,500 calories daily)

Group 2: Follow an intermittent very-low calorie diet (500-800 calories). Participants in this group will alternate between days of 500-800 calories and days of structured eating using healthy eating principles.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years.
2. BMI 25-35. Patients with a BMI less than 25 are not classified as overweight and individuals with a BMI >35 may require more aggressive weight management strategies.
3. Clearance for participation from their PCP.

Exclusion Criteria:

1. Participation in a research project or formal program involving weight loss or exercise in the previous 6 mos., as these proximal experiences may impact the results of this study.
2. Participation in a regular exercise program (i.e., > 500 kcal/wk. of planned activity as estimated by questionnaire [34].
3. Not weight stable (-/+ 5%) for 6 mos. prior to intake. This will be determined by phone screen and self-report on the health history questionnaire
4. Unwilling to be randomized to one of two diet strategies for weight loss.
5. Pregnant during the previous 6 mos., lactating, or planned pregnancy in the following 6 mos.
6. Serious medical risk (e.g. diabetes, cancer, cardiovascular disease) as determined by the individual's physician via the clearance to participate in the investigation.
7. Disordered eating as determined by the Eating Attitudes Test using a score of 20 or greater [35]. This score indicates the need for counseling outside the scope of this study.
8. Current treatment for psychological problems, or taking psychotropic medications. Addressing psychological problems is outside the scope of this study.
9. Medications known to significantly influence weight.
10. Adherence to specialized diet regimens (e.g., multiple food allergies, vegan, etc.)
11. Do not have access to or independence over grocery shopping and meal preparation (i.e. those in military, college with cafeteria plan, etc.).
12. If participants have recently undergone CT (Computed Tomography), PET, fluoroscopic, or nuclear medicine studies within the past year.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Weight (lbs, % change from baseline) | Change from baseline to 24 weeks
  Change in absolute (lbs) and relative (%) weight from baseline to the end of the intervention (24 weeks)
Body composition | Change from baseline to 24 weeks
  Change in absolute (g) and relative (%) fat mass and fat-free mass from baseline to 24 weeks

SECONDARY OUTCOMES:
Program adherence | weekly through study completion (24 weeks)
  Compliance to intervention protocol; adherence = (# attained / # expected)*100
Nutrition-related quality of life | baseline, week 12, week 24
  Assessed via questionnaire; higher scores indicate greater nutrition-related quality of life.
Dietary restraint | baseline, week 12, week 24
  Assessed via three-factor eating questionnaire with three component scores for cognitive restraint, disinhibition, hunger)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Sullivan, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided